CLINICAL TRIAL: NCT02215122
Title: A Bioequivalence Study to Assess the Systemic Exposure of Fluticasone Propionate and Salmeterol Administered as a Fixed Dose Combination From Different Dry Powder Inhalers in Healthy Subjects
Brief Title: Bioequivalence Study to Assess Systemic Exposure of FP and SAL FDC From Different DPIs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharma UK Ltd. (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MGR001-1008
Record Dates: First submitted 2014-08-05; First posted 2014-08-13 (Estimated); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Asthma; COPD
Keywords: Fluticasone Propionate; Salmeterol; Pharmacokinetics; Healthy Subjects; MGR001; CRC749; Dry Powder Inhaler; generic; Advair Diskus; Seretide Accuhaler
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MGR001 (Experimental): FP/SAL 250/50 µg 3 x inhalations (total dose 750/150 µg) administered via CRC749 inhaler.
  Interventions: Drug: MGR001
- Advair® Diskus® (Experimental): FP/SAL 250/50 µg 3 x inhalations (total dose 750/150 µg) administered via Diskus® inhaler.
  Interventions: Drug: Advair® Diskus®
- Seretide™ Accuhaler™ (Experimental): FP/SAL 250/50 µg 3 x inhalations (total dose 750/150 µg) administered via Accuhaler™ inhaler.
  Interventions: Drug: Seretide™ Accuhaler™

INTERVENTIONS:
Drug: MGR001 — Fluticasone Propionate is an inhaled corticosteroid (ICS) Salmeterol is a long acting β2 agonist (LABA)
  Other Names: FP; SAL
  Arms: MGR001
Drug: Advair® Diskus® — Fluticasone Propionate is an inhaled corticosteroid (ICS) Salmeterol is a long acting β2 agonist (LABA)
  Other Names: FP; SAL
  Arms: Advair® Diskus®
Drug: Seretide™ Accuhaler™ — Fluticasone Propionate is an inhaled corticosteroid (ICS) Salmeterol is a long acting β2 agonist (LABA)
  Other Names: FP; SAL
  Arms: Seretide™ Accuhaler™

SUMMARY:
This is a crossover study to assess the systemic pharmacokinetics of fluticasone propionate (FP) and salmeterol (SAL). Study medication will be administered as fixed dose combinations (250 µg FP and 50 µg SAL) from the Advair® Diskus®, Seretide™ Accuhaler™ and CRC749 inhalers.

DETAILED DESCRIPTION:
Study drug will be administered through the inhaled route to healthy subjects in single doses (three inhalations, i.e. total dose 750 µg FP and 150 µg SAL).

Each subject will receive the following treatments in a random order:

A. MGR001 B. Seretide™ Accuhaler™ C. Advair® Diskus® There will be a wash out of 3 7 days between treatment periods. Pharmacokinetics will be assessed by the measurement of plasma concentrations of FP and SAL over the 48 hours following dosing. Adverse Events will be collected throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years.
* Body Mass Index (BMI) of 18 to 30.5 kg/m2; and a total body weight >45 kg (99 lbs).
* An informed consent document signed and dated by the subject.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 14 units/week for females or 21 units/week for males (1 unit = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
* Treatment with an investigational drug within 30 days or 5 half-lives or as determined by the local requirement, whichever is longer, preceding the first dose of study medication.
* 12-lead ECG demonstrating QTcF >450 msec or a QRS interval >120 msec at screening. If QTcF exceeds 450 msec or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTcF or QRS values should be used to determine the subject's eligibility.
* Hemoglobin <11.5 g/dL for female subjects or <12.5 g/dL for male subjects.
* Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of contraception as outlined in this protocol.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study medication. Herbal supplements must be discontinued at least 28 days prior to the first dose of study medication. - Blood donation of approximately 1 pint (500 mL) or more within 56 days prior to dosing.
* Unwilling or unable to comply with the lifestyle guidelines described in this protocol.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results.
* Evidence or significant history of childhood or adult asthma, or any significant history of wheeze, chronic cough, dyspnea at rest or acute bronchospasm.
* Subjects with abnormal lung function tests at screening, defined as an FEV1 and/or FVC which is <80% of predicted.
* Subjects who are current smokers. Ex-smokers who have given up smoking for <6 months and/or have a smoking pack history of ≥10 pack years.
* Subjects with a lower respiratory tract infection in the 4 weeks prior to dosing.
* History of sensitivity to lactose or sensitivity to the ingredients of Advair®/Seretide™, including subjects with severe milk protein allergy in whom Advair® is contraindicated.
* Subject is the Investigator or a sub-Investigator, research assistant, pharmacist, study coordinator, other staff, or a relative of any study personnel directly involved with the conduct of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
AUC for each of the treatment groups FP/SAL | 3 days of each treatment period.
Cmax for each of the treatment groups FP/SAL, | 3 days of each treatment period.

SECONDARY OUTCOMES:
Adverse events | Day1 to Day3
Inspiratory Flow assessments | Day 1 pre-dose

CONTACTS AND LOCATIONS:
Overall Officials: Jon Ward, Study Director — Mylan Pharma UK Ltd.
Locations (1):
- Worldwide Clinical Trials Early Phase Services, San Antonio, Texas, United States